CLINICAL TRIAL: NCT05859139
Title: PEGASUS-2: Scaling a Decision Aid on Prenatal Screening for Trisomy 21, 18 and 13: A Stepped Wedge Cluster Randomized Trial
Brief Title: Scaling a Decision Aid on Prenatal Screening for Trisomy 21, 18 and 13
Acronym: PEGASUS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, France Legare, Professor, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: MP-13-2022-2574
Record Dates: First submitted 2023-03-29; First posted 2023-05-15 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Decision Aid
Keywords: Decision Aid; Health Professionals; Scaling strategies; Online training; Prenatal screening; Shared decision-making; Trisomy; Pregnant women; Prenatal services
MeSH Terms: conditions — Trisomy

STUDY DESIGN:
Intervention Model Description: This study will consist of four groups receiving the intervention in a sequential way. Each group will include several prenatal services corresponding to the study clusters (the randomization unit). Randomization will occur at the site level. Clinics will be randomized in groups to receive the intervention. At the end, every clinic will be in intervention conditions. The study will be conducted over five periods each corresponding to a data collection period. During the first period, all groups will be in control conditions where health professionals will provide the usual prenatal care to pregnant women (no intervention). Then, after a regular interval of 10 weeks, each group will receive the intervention starting with the beginning of the remaining four periods. Once a group has received the intervention, it will remain in intervention conditions until the end of the study.
Who Masked: Outcomes Assessor
Masking Description: Allocation of prenatal services to groups and stages will be blinded by an independent, experienced biostatistician who will not be involved in the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention introduced to group 1 (Experimental): The intervention is introduced to the first group (G1) of clusters.
  Interventions: Other: DA Scaling Strategies
- Intervention introduced to group 2 (Experimental): The intervention is introduced to the second group (G2) of clusters and G1 remains in intervention conditions.
  Interventions: Other: DA Scaling Strategies
- Intervention introduced to group 3 (Experimental): The intervention is introduced to the third group (G3) of clusters and G1 and G2 remains in intervention conditions.
  Interventions: Other: DA Scaling Strategies
- Intervention introduced to group 4 (Experimental): The intervention is introduced to the fourth group (G4) of clusters and G1, G2 and G3 remains in intervention conditions.
  Interventions: Other: DA Scaling Strategies

INTERVENTIONS:
Other: DA Scaling Strategies — For this study the intervention will consist of different DA scaling strategies : 1) dissemination of an online DA; 2) dissemination of a paper-based DA; 3) online training for healthcare professionals.

SUMMARY:
This research project aims at assessing the effectiveness of a decision aid (DA) scaling intervention within the context of prenatal screening for trisomy 21, 18 and 13. The primary outcome is the level of involvement of pregnant women, their partners, and health professionals in shared decision-making (SDM) in the context of prenatal screening for trisomy 21, 18 and 13. The secondary outcome is the rate of use of online and paper versions of the DA by pregnant women, their partners and health professionals. The investigator hypothesize that the DA scaling strategies will increase the level of involvement of pregnant women, their partners (where appropriate), and health professionals in SDM.

DETAILED DESCRIPTION:
Making a decision about prenatal screening for trisomy 21, 18 and 13 can be difficult. This is why it is important for pregnant women and their partners to be informed, accompanied and supported by health care providers. Involving them in shared decision-making (SDM) would allow them to meet their decision-making needs in this context. In addition, the use of a decision aid (DA) would facilitate SDM. To help pregnant women and their partners make informed decisions based on their values, needs and preferences, a DA has been developed. The DA was developed according to recommendations from pregnant women and their partners as well as health professionals who found it relevant. Moreover, the DA scaling up strategies were developed. This research project aim is to assess the effectiveness of the DA scaling strategies on the level of involvement of pregnant women, their partners, and health professionals in SDM on prenatal screening for trisomy 21, 18 and 13. This study, conducted in Quebec, is a randomized cluster stepped wedge trial. The study will be conducted in five periods, each corresponding to a data collection period. During the first period, all groups of clusters will be in control conditions, where health professionals will provide usual prenatal care to pregnant women without DA scaling strategies. Then, following a regular interval of 10 weeks, each group will be exposed to the intervention in 4 stages at the beginning of the periods. Once a group has received the intervention, they will access it until the end of the study. Participants are prenatal services (randomization unit), health professionals (obstetricians-gynecologists, family physicians, midwives, nurses and all other health professionals involved in prenatal care) and pregnant women as well as their partners. The intervention will consist of a DA scaling strategies, including but not limited to an online version of the DA and an online training on SDM incorporating the use of the DA. The investigators will recruit at least 28 prenatal services (study sites) and 35 pregnant women per site. The primary outcome (the level of involvement of study participants in SDM in the context of prenatal screening for trisomy 21, 18 and 13) will be measured with the validated SDM-Q-9 scale, which will be completed by pregnant women and their partners. The primary secondary outcome will be the rate of use of online and paper versions of the DA by pregnant women and their partners.

ELIGIBILITY:
Inclusion Criteria:

• Prenatal services (study sites) : To be eligible, prenatal services must

* be located in Quebec province
* be family medicine groups, gynecology and obstetrics departments or birth centers, other type of health facility involved in prenatal care
* agree to participate in our study including the recruitment of approximately 35 pregnant women over a total period of 50 weeks
* confirm that they will follow the research protocol.

  * Health professionals

To be eligible, health professionals must:

* be involved in prenatal care and working in a site participating in this study
* be involved in the follow-up of pregnancies
* be involved in the decision-making process in the context of prenatal screening for trisomiy 21, 18 and 13,
* be referred by their prenatal service
* understand French or English,
* consent to participate in the study
* medical residents and interns in midwifery practice, referred by participating prenatal service, are eligible too.

  • Pregnant women and their partners To be eligible, pregnant women and their partners must
* be 18 years of age or older
* have not yet decided whether or not to have prenatal testing for trisomy 21, 18 or 13 (usually before 13 weeks of pregnancy)
* be followed in one of the prenatal services participating in this study
* be able to read and understand French or English
* have the capacity to verbally consent to participate in the study or sign the consent form

Exclusion Criteria:

* Pregnant women and their partners The pregnant woman who have any medical complications associated or not with pregnancy (e.g. diabetes, hypertension, multiple pregnancy) is not eligible to this study
* Health professionals Health professionals working in more than one participating prenatal site as full- time or part-time employee are not eligible to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 887 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Level of SDM adoption | At the 23rd week of pregnancy
  The level of SDM adoption will be measured through the measurement of the level of involvement of health professionals and pregnant women (and their partners) in the decision regarding to have or not a prenatal screening test for trisomy 21, 18 and 13. The SDM adoption will be measured with the SDM-Q-9 scale, which is a validated measurement instrument. The SDM-Q-9 scale is well understood by patients and has the potential to collect valid data on the perceived involvement of patients in SDM. The SDM-Q-9 scale consists of 9 items, each corresponding to the expected behaviour of the health professional in the SDM. Each of the 9 items is rated by a six-point Likert scale (0 = Totally Disagree to 5 = Totally Agree) where higher scores reflect higher level of SDM adoption.

SECONDARY OUTCOMES:
The rate of the DA utilization by pregnant women, their partners and health professionals | At the 23rd week of pregnancy (for pregnant women and their partners), and the research team will compile the information on the online and hard copies of DA utilization during weeks 10 to 50 of the study (Intervention phases)
  At the 23rd week of pregnancy, pregnant women and their partners will answer questions about whether they used the DA to help them make their decision. For each intervention period of the study, the research team will compile the number of utilization of the online DA as well as the city of the users. The research team will also track the number of hard copies of the DA used by each prenatal service recruited.
Perceived role in decision-making | At the 23rd week of pregnancy
  Pregnant women and their partners will be be asked to assess their perceived role in deciding whether or not to have prenatal screening for trisomies 21, 18 and 13. The investigators will use a validated 1-question scale with five options of responses (A, B, C, D and E). The investigators will combine choices A and B to identify the proportion of pregnant women (and their partners) who will have made the decision alone, choice C to identify the frequency of SDM, and thte investigators will combine D and E choices to identify the proportion of pregnant women (and their partners) who have had a passive role.
DA appreciation | At the 23rd week of pregnancy
  This study will assess the participants' general appreciation of the DA. Once pregnant women and their partners have used the online or paper DA, they will respond to a questionnaire (questions with different options of responses) assessing their appreciation on the DA (on its presentation, acceptability, usefulness, neutrality, quantity and quality of information, etc.). Questions to be responded to will be adapted according to the version used (online or paper based DA).
Appreciation of the online SDM training | Immediately after the online training
  Once health care professionals have completed the online SDM training, they will respond to questions aiming at assessing their overall appreciation (on its presentation, acceptability, usefulness, quantity and quality of information, etc.). Open-ended questions will allow them to say what they liked or did not like, to offer suggestions for improvement or to add any other comments.
Decisional conflict | At the 23rd week of pregnancy
  To measure the level of decisional conflict among pregnant women and their partners, the investigators will use the validated scale that assess the decisional conflict. The scale has 16 items evaluated with a 5-point Likert scale (1 = Strongly agree, 5 = Strongly disagree).
Decisions made and chosen tests | At the 23rd week of pregnancy
  Pregnant women and their partners will answer questions about what was their decision as to whether or not to do a screening test. If they chose to do a screening test, what was the test(s) and whether the test(s) was done in the public or private network. In addition, they will be asked if they went further for a diagnostic test.
Facilitators and barriers to the use of the DA | At the 23rd week of pregnancy
  Pregnant women and their partners will be asked open-ended questions to find out what helped, or allowed, and what limited, or prevented them from using our DA in the format used (paper based or online DA).
Duration of the prenatal consultation | At the 23rd week of pregnancy
  The investigators will ask pregnant women and their partners how long the targeted prenatal consultation (with the discussion on prenatal testing ) lasted.
Efforts and costs related to the use of the DA | At the 23rd week of pregnancy
  Pregnant women and their partners will answer questions about whether they used our DA, and if so, will follow questions aiming at assessing the energy or effort invested in using it and the possibility that the use of the DA was associated with financial expenses or losses.
Efforts and costs related to the use and the distribution of the DA | Immediately after the intervention
  The investigators will ask prenatal service leaders or champions what level of effort and energy they had to invest to use and/or distribute the DA to pregnant women and their partners. In addition, the investigators will ask them if the use and/or distribution of the DA caused them financial expenses or losses, or if this required more human resources.
DA use fidelity for pregnant women and their partners | At the 23rd week of pregnancy
  After deciding whether to do or not the prenatal screening test, pregnant women and their partners will answer questions to assess the extent to which they have used the tool (e.g. number of sections read and/or completed) and when they used it. These questions are used to assess whether pregnant women (and their partners) used the tool as intended.
DA use fidelity for healthcare providers | At the 23rd week of pregnancy
  A set of questions will be asked to pregnant women and their partners to assess whether a person has given them the DA (in hard copy or the internet link), and if so, by whom and when. The investigators also want to know if the healthcare providers used the DA during the prenatal consultation and how.
Long-term use of DA and proposed adaptations for the DA | At the 23rd week of pregnancy
  Pregnant women and their partners will answer questions to assess whether they intend to reuse the DA for a future pregnancy or if they would like to use another DA for another medical decision.

CONTACTS AND LOCATIONS:
Overall Officials: France Légaré, Ph.D, Principal Investigator — Laval University
Locations (1):
- VITAM - Centre de recherche en santé durable, CIUSSS de la Capitale-Nationale, Québec, Canada

REFERENCES:
- See also: Related Info — http://www.decision.chaire.fmed.ulaval.ca/